CLINICAL TRIAL: NCT05064163
Title: Social Return on Investment (SROI) Project of the Surgical Waiting List Management System
Brief Title: SROI Project on the Surgical Waiting List Management System
Status: Completed | Type: Observational
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, Jose Luis Gonzalez Munoz, Principal Investigator, University of Malaga
Other Study IDs: SROI-LEQ2020; 113.21 (Registry Identifier: CÁDIZ RESEARCH ETHICS COMMITTEE)
Record Dates: First submitted 2021-09-01; First posted 2021-10-01 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Digestive System Disease
Keywords: Social Return on Investment (SROI); Surgical waiting list; Health Concerts; Diagnostic tests; Surgical procedures
MeSH Terms: conditions — Digestive System Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The waiting lists for surgery and diagnostic tests registered in the health management area of Campo de Gibraltar West are very high, and this is compounded by the lack of resources that prevent them from being managed efficiently.

The aim of the study is to know, quantify and communicate the measurement of the social impact, also known as social return on investment, which is presented as a tool for decision making on the intervention of the management of health concerts in comparison with the current system in Andalucia.

In addition, other objectives will be studied, such as the health and non-health benefits derived from applying the intervention of the concerts compared to the current system of waiting list management from the economic, social and environmental points of view, the economic cost of the interventions by the health concerts and the Andalusian public health system, the cost of the increase in extraordinary health resources, determining the most prevalent surgeries from highest to lowest and specifying the highest number of surgeries that are established in the concerts and in the SSPA.

The method used will be an economic evaluation of the different healthcare technologies in which the investigators compare the healthcare agreements of the most prevalent procedures and those that collect data in both groups through the SROI tool. A cross-sectional and prospective design will be carried out with a time horizon of 2021 and 2022, and for the statistical analysis the investigators will use the SSPS V25 and JASP programmes.

The investigators consider it necessary to carry out this research study as there is no specific bibliography on the healthcare technology used in healthcare agreements as a new healthcare technology compared with the current system for managing surgical waiting lists in the Andalusian public healthcare system in terms of return on investment.

DETAILED DESCRIPTION:
The main objective of the study is to carry out a SROI (social return on investment) project as a decision-making tool for clinical and health management of waiting lists in Campo de Gibraltar.

In addition, the investigators consider it necessary to carry out this research study as there is no specific bibliography on the healthcare want to achieve other more specific objectives such as:

* To know the economic cost of the interventions by the extraordinary health concert and the ordinary activity of the Andalusian Public Health System (APHS) of the surgical waiting list and diagnostic tests of certain surgical and functional procedures.
* To know the increase in extraordinary resources to reduce waiting lists in terms of human and material resources.
* To describe socio-demographic data and the prevalence of surgical interventions and diagnostic tests in the extraordinary agreement and the Andalusian Public Health System (APHS).
* To find out how the patient's life is affected in different areas.
* Specify the patient's willingness to pay to improve their quality of life.
* To determine the social return for each surgical procedure and functional test.

The methodology of the study, a questionnaire will be carried out with the aim of analysing the effect that the waiting list for surgery and diagnostic tests has on the lives of the people who suffer from it, this questionnaire will include, among others, the following sections:

* Socio-demographic characteristics, employment situation and family environment.
* Type of procedures and pathology - Effect of the waiting list for surgery and diagnostic tests on different areas of the patient's life.
* Willingness to pay to improve aspects of their life affected since diagnosis.
* Use of health resources in the last year linked to the pathology.

The number of visits that the patient will have to make will only be once, prior to their diagnostic or surgical procedure, to which they will be given the information sheet, informed consent and questionnaires.

Extraordinary visits will not be made. The alternative procedures or treatments that may exist for the subject and their significant potential risks and benefits.

The duration of the study will be 1 year, from April 2021 to March 2022. The number of participants will be the patients included in the surgical waiting list and diagnostic tests of the Hospital Punta de Europa located in the health management area Campo de Gibraltar West and referred to the centre "Clínica Virgen del Rosario".

ELIGIBILITY:
Inclusion criteria:

* Patients undergoing surgery and diagnostic tests at Hospital Punta Europa in ordinary activity.
* Patients undergoing surgery and diagnostic tests in external health care agreement at the Clínica Virgen del Rosario in Algeciras.

Exclusion criteria:

* Urgent surgical interventions -Urgent diagnostic tests.
* Patients who have signed the revocation of informed consent.
* Absence at the surgical appointment - Lack of collaboration
* Resolution of the illness causing the surgical appointment. No presentation of illness
* Refusal by the physician
* Allergies

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients on the waiting list for surgery and diagnostic tests at the Hospital Punta de Europa, located in the Campo de Gibraltar West health management area, and referred to the "Clínica Virgen del Rosario" centre.
Sampling Method: Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-05-16 (Actual)

PRIMARY OUTCOMES:
Economic cost | 4 months
  To ascertain the economic cost of interventions under the extraordinary healthcare agreement and of the ordinary activity of the Andalusian Public Health System (APHS) of the surgical waiting list and of diagnostic tests for certain surgical and functional procedures.
Increase in resources | 4 months
  To know the increase in extraordinary resources to change waiting lists in terms of human and material resources.
Prevalence of surgical procedures | 4 months
  Calculate by dividing the total number of individuals with a surgical procedure at the time of the study by the population at that point in time.
Quality-adjusted life years (QALYs) | 4 months
  Determine QALYs by multiplying the utility value associated with a given health state by the years lived in that state.
Rate of return on investment (SROI) | 4 months
  Determine the social return for each surgical procedure and functional test.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Virgen Del Rosario, Algeciras, Cadiz, Spain

DOCUMENTS (1):
  • Informed Consent Form (2021-07-12): https://cdn.clinicaltrials.gov/large-docs/63/NCT05064163/ICF_000.pdf